CLINICAL TRIAL: NCT06296368
Title: DISCOVERY: Evaluating a Decision Support Tool for Adults Seen in Hematology/Oncology Clinics
Acronym: DISCOVERY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LCCC2305; K08CA273684-01A1 (NIH)
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Malignancies; Lymphoma; Multiple Myeloma; Leukemia; Blood Cancers
Keywords: decision support tool; pragmatic study; best-worst scaling
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Receive usual care.
- PRIME intervention (Experimental): Receive the PRIME intervention.
  Interventions: Behavioral: Preference Reporting to Improve Management and Experience (PRIME)

INTERVENTIONS:
Behavioral: Preference Reporting to Improve Management and Experience (PRIME) — PRIME is a decision support tool that uses best-worst scaling to provide a personalized report to providers and patients of their most important treatment priorities
  Arms: PRIME intervention

SUMMARY:
The purpose of this study is to evaluate whether a novel decision support tool called PRIME (Preference Reporting to Improve Management and Experience), which combines values-elicitation with tailored feedback to patients and providers, improves patient-reported values-concordance of initial treatment decisions compared to usual care.

DETAILED DESCRIPTION:
In the last decade, remarkable advances in drug development have led to the approval of 52 new therapies for patients with hematologic malignancies. These new approvals are increasingly enabling clinicians to personalize chemotherapy decisions to achieve what matters most to patients. Therefore, accurately assessing patient preferences is critical to personalizing treatment decisions, particularly among older adults, who face high treatment-related morbidity and/or shorter anticipated survival.

Patient preferences have traditionally been inferred from face-to-face conversations. However, numerous studies, including several systematic reviews, have demonstrated that this process alone is inadequate to reliably capture patient preferences. To support standard shared decision making, multiple stakeholders strongly advocate the development of validated patient-reported measures that accurately capture patients' preferences. In recent guidance about the care of older adults with leukemia, the American Society of Hematology explicitly recommends the development of novel decision support tools to address this growing challenge in patient-centered care. Improved shared decision making has been associated with increased patient-reported quality of care and satisfaction, and a reduction in healthcare utilization.

This study will determine the effectiveness of a novel decision support tool called "PRIME" (Preference Reporting to Improve Management and Experience) to improve the values-concordance of initial treatment decisions. Using best-worst scaling, a validated values-elicitation method, PRIME provides a personalized report to providers and patients of their most important treatment priorities.

In this pragmatic trial, participants will be randomized to receive decision support with PRIME or usual care prior to their first visit with their oncologist. The primary outcome will be clinically significant improvement in values-concordance of the initial treatment decision (on CollaboRATE, a validated 12-point measure).

ELIGIBILITY:
Inclusion Criteria In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

1. Written or verbal informed consent obtained to participate in the study and HIPAA authorization for the release of personal health information.
2. Subjects are willing and able to comply with study procedures based on the judgment of the investigator.
3. Age ≥ 60 years at the time of consent.
4. New patient to either the hematologic malignancies clinic or the bone marrow transplant/cellular therapy clinic.

Exclusion Criteria

All subjects meeting any of the exclusion criteria listed below at baseline will be excluded from study participation:

1. Dementia, altered mental status, or psychiatric condition that would prohibit the understanding or rendering of informed consent or participation in the intervention.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in COLLABORATE scores between arms | Up to 24 months
  The effectiveness of PRIME to improve the value-concordance of treatment decisions in older subjects presenting to hematologic malignancy clinics will be determined by differences in CollaboRATE scores (Percentage in each arm that report perfect scores 15/15) at the post-treatment decision assessment between control and intervention groups.
  COLLABORATE scores is a Likert scale questionnaire that includes 3 questions rated from 1 to 5. Higher scores represent better patient engagement.

SECONDARY OUTCOMES:
Difference in COLLABORATE scores between arms in a subgroup of patients | Up to 24 months
  The secondary outcome will be the difference in CollaboRATE scores (percentage in each arm that report perfect scores 15/15) at the post-treatment decision assessment between control and intervention groups in a subgroup of participants: participants with newly-diagnosed Acute myeloid leukemia, Acute Lymphoblastic leukemia, Diffuse Large B-cell Lymphoma, and Multiple myeloma COLLABORATE scores is a Likert scale questionnaire that includes 3 questions rated from 1 to 5. Higher scores represent better patient engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Richardson, MD, MA, MSc, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comphrehensive Cancer Center at University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials